CLINICAL TRIAL: NCT07114133
Title: A Study on the Efficacy of Environmental Probiotics in Patients With Cat Hair Allergies
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2025-0723
Record Dates: First submitted 2025-07-20; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-07

CONDITIONS: Cat Allergy (Disorder); Allergic Rhinitis; Allergic Asthma
Keywords: Cat Allergy; Allergic Rhinitis; Allergic Asthma; Environmental Probiotics
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Environmental Probiotic Spray Intervention Arm (Experimental): Participants in this arm will administer the environmental probiotic spray at home according to the following protocol:
  First bottle: 3 times daily (TID), 30 actuations per administration Subsequent bottles (from second bottle onward): Once daily (QD), 15 actuations per administration Total duration: 3 months
  Interventions: Other: Environmental Probiotic Spray Intervention
- Purified Water Spray Intervention Arm (Placebo Comparator): Participants in this arm will administer the purified water spray at home according to the following protocol:
  First bottle: 3 times daily (TID), 30 actuations per administration Subsequent bottles (from second bottle onward): Once daily (QD), 15 actuations per administration Total duration: 3 months
  Interventions: Other: Purified water spray (containing no active ingredients) as the placebo control

INTERVENTIONS:
Other: Environmental Probiotic Spray Intervention — The probiotic strains include Bacillus subtilis YHX001J, Bacillus amyloliquefaciens YHX002J, and Bacillus velezensis YHX003J
  Arms: Environmental Probiotic Spray Intervention Arm
Other: Purified water spray (containing no active ingredients) as the placebo control — Purified water spray
  Arms: Purified Water Spray Intervention Arm

SUMMARY:
Objective of this clinical trial:

The goal of this clinical study is to evaluate whether an environmental probiotic spray can improve symptoms in adults with cat allergy-induced allergic rhinitis (AR) and allergic asthma (AA). It will also assess the safety of the probiotic spray. The main questions it aims to answer are:

Does the environmental probiotic spray reduce the severity of nasal and asthma symptoms in participants? Are there any adverse effects observed in participants using the probiotic spray? Researchers will compare the environmental probiotic spray group to a placebo group (a look-alike spray containing no active ingredients) to determine if the probiotic spray is effective in managing allergic rhinitis and asthma symptoms.

Participants will:

Receive the environmental probiotic spray or placebo daily for 3 months Attend monthly clinic visits for checkups and assessments Undergo a final evaluation at 3 months, including symptom scoring and safety checks

Key Assessments:

Total Nasal Symptom Score (TNSS) for allergic rhinitis Asthma Control Test (ACT) score for allergic asthma

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years；
* Diagnosed with cat allergy (cat dander-specific IgE level ≥ class 2: > 0.7 IU/mL) and allergic rhinitis with or without allergic asthma;
* Residing in the same living environment for at least 3 months (and no plans to change residence within the next 6 months);
* Patients receiving conventional symptomatic treatment.

Exclusion Criteria:

* Presence of other severe systemic diseases;
* Residence duration < 3 months or plans to change residence within the next 6 months;
* Pregnancy;
* Current or planned use of biologic therapy;
* Any other condition that, in the investigator's judgment, may pose significant risks to the participant if enrolled in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the TNSS score at 3 Months | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No